CLINICAL TRIAL: NCT03038568
Title: Stability of Radiomic Features for Abdominal Tumors on Contrast Enhanced CT
Brief Title: Assessing How Normal Variations in CT Scanning Affects Its Interpretation
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Kingston Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 17-010
Record Dates: First submitted 2017-01-30; First posted 2017-01-31 (Estimated); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer Metastatic
Keywords: colorectal liver metastases; CT scan; 17-010
MeSH Terms: interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (18):
- Cohort 1: -15 second time gap between routine abdominal CT and add on CT, Noise Index of 12
  Interventions: Diagnostic Test: CT scan
- Cohort 2: -15 second time gap between routine abdominal CT and add on CT, Noise Index of 14
  Interventions: Diagnostic Test: CT scan
- Cohort 3: -15 second time gap between routine abdominal CT and add on CT, Noise Index of 16
  Interventions: Diagnostic Test: CT scan
- Cohort 4: -10 second time gap between routine abdominal CT and add on CT, Noise index 12
  Interventions: Diagnostic Test: CT scan
- Cohort 5: -10 second time gap between routine abdominal CT and add on CT, Noise index 14
  Interventions: Diagnostic Test: CT scan
- Cohort 6: -10 second time gap between routine abdominal CT and add on CT, Noise index 16
  Interventions: Diagnostic Test: CT scan
- Cohort 7: - 5 second time gap between routine abdominal CT and add on CT, Noise index 12
  Interventions: Diagnostic Test: CT scan
- Cohort 8: - 5 second time gap between routine abdominal CT and add on CT, Noise index 14
  Interventions: Diagnostic Test: CT scan
- Cohort 9: - 5 second time gap between routine abdominal CT and add on CT, Noise index 16
  Interventions: Diagnostic Test: CT scan
- Cohort 10: + 5 second time gap between routine abdominal CT and add on CT, Noise index 12
  Interventions: Diagnostic Test: CT scan
- Cohort 11: + 5 second time gap between routine abdominal CT and add on CT, Noise index 14
  Interventions: Diagnostic Test: CT scan
- Cohort 12: + 5 second time gap between routine abdominal CT and add on CT, Noise index 16
  Interventions: Diagnostic Test: CT scan
- Cohort 13: + 10 second time gap between routine abdominal CT and add on CT, Noise index 12
  Interventions: Diagnostic Test: CT scan
- Cohort 14: + 10 second time gap between routine abdominal CT and add on CT, Noise index 14
  Interventions: Diagnostic Test: CT scan
- Cohort 15: + 10 second time gap between routine abdominal CT and add on CT, Noise index 16
  Interventions: Diagnostic Test: CT scan
- Cohort 16: + 15 second time gap between routine abdominal CT and add on CT, Noise 12
  Interventions: Diagnostic Test: CT scan
- Cohort 17: + 15 second time gap between routine abdominal CT and add on CT, Noise 14
  Interventions: Diagnostic Test: CT scan
- Cohort 18: + 15 second time gap between routine abdominal CT and add on CT, Noise 16
  Interventions: Diagnostic Test: CT scan

INTERVENTIONS:
Diagnostic Test: CT scan — Patients with colorectal liver metastases scheduled for abdominopelvic CECT will be consented to undergo an additional CT of their abdomen (termed add-on CT) within 15 seconds, before or after, their clinical portal venous phase CT (PV CT), which is performed at a fixed delay of 80 seconds at our institution.

SUMMARY:
The purpose of the study is to see how measurements of tumor differences vary with slight changes in CT scan parameters. Reproducible radiomic features can be extracted for abdominal tumors, and specifically colorectal liver metastases, imaged with clinical CT scanners even in the setting of variable scan parameters and variable contrast timing. Participants will be consented to undergo an additional CT of their abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age on the day of signed informed consent
* Patients scheduled and approved for contrast enhanced CT that includes imaging of the abdomen and pelvis following the Department of Radiology standard of care protocol as per local institutional guidelines
* Patients with measurable colorectal liver metastases on prior imaging, with at least one tumor greater than 2.0 cm in axial maximal diameter

Exclusion Criteria:

* Patient who is pregnant and/or lactating
* Patient scheduled for CT that includes the abdomen with a multiphasic contrast enhanced protocol (e.g. Triple Phase or Quadruple Phase Liver CT)
* Patient who require reduced intravenous contrast dose based on the Department of Radiology contrast policy as per local institutional guidelines
* Any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or follow up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo contrast enhanced CT scanning for colorectal liver metastases will be consented for one additional CT abdomen phase during the same imaging session.
Sampling Method: Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2026-01-27 (Estimated); Study Completion 2026-01-27 (Estimated)

PRIMARY OUTCOMES:
assess the stability (reproducibility) of radiomic measurements obtained from repeat abdominal CT scans | 2 years
  There will be 18 cohorts, each cohort differing by the length of the time gap in acquisition and noise index. In addition each acquisition will be reconstructed in 21 different ways (combinations of 3 slice thicknesses and 7 ASiR levels).

CONTACTS AND LOCATIONS:
Overall Officials: Kinh Gian Richard Do, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Texas (Data collection only), Houston, Texas

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

DOCUMENTS (1):
  • Informed Consent Form (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/68/NCT03038568/ICF_000.pdf